CLINICAL TRIAL: NCT00230906
Title: Uremic Toxin Removal With a New High Flux Cellulose Triacetate Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Nissho Nipro Europe (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2001/182
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Haemodialysis
MeSH Terms: interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Haemodialysis with either low or high flux membranes

SUMMARY:
Comparison of the uremic toxin removal by haemodialysis either with a low flux or a new high flux cellulose triacetate membrane

DETAILED DESCRIPTION:
Comparison of the uremic toxin removal by haemodialysis either with a low flux or a new high flux cellulose triacetate membrane

ELIGIBILITY:
Inclusion Criteria:

* Chronic haemodialysis patient
* Serum albumin > 3.6 g/dl

Exclusion Criteria:

* < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2001-01; Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Concentration of uremic components after 3 weeks of haemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Van Holder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be